CLINICAL TRIAL: NCT03791411
Title: Narratives and Reflective Practice: A Programme for the Development of Professional Competences in Nursing
Brief Title: Nursing Narratives, Reflective Practice and Professional Development (NarratUN)
Acronym: NarratUN
Status: Completed | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: NPR
Record Dates: First submitted 2018-12-21; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-04

CONDITIONS: Narrative Medicine
Keywords: Clinical Narratives; Respect; Intentional presence; knowing the person; Professional development
MeSH Terms: conditions — Narrative Medicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: In addition to foster reflective practice, clinical narratives may be used as a means to improve nurses' critical thinking and their acquisition of clinical competencies. However, few studies have studied their potential value to promote nursing professional development and there is no evidence that shows their value as a tool to improve nurses' competencies to provide a person-centred nursing care.

Purpose: To evaluate the preliminary efficacy of narratives for the development of three nursing professional competences -respect, intentional presence and knowing the person- paramount to provide person-centred care.

Method: A pilot quasi-experimental study. A total of 34 nurses enrolled in a global training course of a nursing specialization were recruited in September 2016. All the nurses received a multi-component intervention based on the Critical Reflexive Inquiry Model. The strategies of this program consisted in the writing of 3 narratives; 3 masterclass of 3, 2 and 3 hours respectively; a discussion group; and a face-to-face interview. The NarratUN Evaluation tool was used to assess outcomes. The primary outcome was the difference in the mean of respect, intentional presence and knowing the person pre and post intervention. Changes within nurses were analyzed using Wilcoxon signed Rank test.

ELIGIBILITY:
Inclusion Criteria:

* Being in a specialized training programme

Exclusion Criteria:

* Not being in a specialized training programme

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nurses enrolled in a global training course of nursing specialization, for the 2016-17, 2017-18, and 2018-19 courses. All students in the specialized training programme will be included, regardless of age or previous experience.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Respect. Measurement tool: NarratUN Evaluation Tool (NET) | 9 month
  The difference in the mean of respect value (pre-post)
Intentional presence. Measurement tool: NarratUN Evaluation Tool (NET) | 9 month
  The difference in the mean of intentional presence value (pre-post)
Knowing the person. Measurement tool: NarratUN Evaluation Tool (NET) | 9 month
  The difference in the mean of knowing the person value (pre-post)

SECONDARY OUTCOMES:
Handling the narrative. Measurement tool: NarratUN Evaluation Tool (NET) | 9 month
  The difference in the mean of Handling the narrative value (pre-post)
Respect. Measurement tool: NarratUN Evaluation Tool (NET) | 2 month follow-up
  The difference in the mean of respect value along different times of the study
Intentional presence. Measurement tool: NarratUN Evaluation Tool (NET) | 2 month follow-up
  The difference in the mean of intentional presence value along different times of the study
Knowing the person. Measurement tool: NarratUN Evaluation Tool (NET) | 2 month follow-up
  The difference in the mean of knowing the person value along different times of the study
Handling the narrative. Measurement tool: NarratUN Evaluation Tool (NET) | 2 month follow-up
  The difference in the mean of Handling the narrative value along different times of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Ana Choperena Armendáriz, Pamplona, Navarre, Spain